CLINICAL TRIAL: NCT07376733
Title: Efficacy of a Controlled Breathing and Therapeutic Exercise Program on Cardiorespiratory Variables in Patients With Multiple Myeloma
Brief Title: Effects of Controlled Breathing on Cardiorespiratory Variables in Multiple Myeloma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Isidro Fernández López, Principal Investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Cardiorespiratory Mieloma
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma (MM); Breathing Techniques; Breathing Exercises; Exercise Activity; Diaphragmatic Breathing; Heart Rate Variability (HRV)
Keywords: multiple myeloma; Breathing; Diaphragmatic breathing; Slow breathing; exercise activity; Breathing exercises; heart rate variability
MeSH Terms: conditions — Multiple Myeloma; Respiratory Aspiration; Hypoventilation | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: A randomized, parallel, double-blind, controlled clinical trial. Two groups of participants will be included, both receiving an educational session with a standardized educational leaflet on the importance of proper breathing, and a therapeutic exercise intervention over a 6-week period. One of the groups will additionally perform a home-based controlled breathing exercise protocol. Pre- and post-intervention assessments (6 weeks) will be conducted, along with a follow-up evaluation 4 weeks after completion of the intervention. For heart rate and heart rate variability variables, two assessments will be conducted at identical time points to determine the immediate within-session effect of the in-person breathing session, compared with participants in the control group, who will be instructed to breathe spontaneously while maintaining their usual breathing pattern.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Only the principal investigator will have access to the randomization sequence, thereby maintaining blinding for the rest of the team involved in data collection. Both groups will receive the same therapeutic exercise program and an educational session with a standardized educational leaflet on the importance of physical activity and proper breathing in daily life, with the aim of minimizing differences in the perceived intervention. The study will include evaluator blinding, as all assessments will be carried out by an independent investigator who is not involved in the randomization process and is unaware of participants' group allocation. Additionally, statistical analyses will be conducted by a specialized statistician, also blinded to group assignment, thereby ensuring impartiality in the analysis and interpretation of the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic exercise + initial education session + home-based controlled breathing exercise protocol (Experimental): * Participants will perform a controlled breathing protocol at home twice daily, at least five days per week, throughout the 6-week study period, following the recommendations of the principal investigator. Additionally, within this same group, two in-person controlled breathing training sessions, each lasting 5 minutes, will be conducted at the hospital.
  * Perform three weekly sessions of mobility and muscle-strengthening exercises (two on-site and one home-based) for 6 weeks. The home-based exercise program will consist of completing, once per week during the 6-week intervention, a structured session that replicates the logic and technique of the on-site program.
  * Walk a minimum of 7,000 steps/day or 50 minutes/day, three days per week.
  * All participants will receive an initial educational session and an explanatory leaflet outlining the fundamental principles of functional breathing.
  Interventions: Other: Controlled breathing exercise protocol + therapeutic exercise + initial education session
- Therapeutic exercise + initial educational session on proper breathing (Active Comparator): * Perform three weekly sessions of mobility and muscle-strengthening exercises (two on-site and one home-based) for 6 weeks. The home-based exercise program will consist of completing, once per week during the 6-week intervention, a structured session that replicates the logic and technique of the on-site program.
  * Walk a minimum of 7,000 steps/day or 50 minutes/day, three days per week.
  * To promote adherence to the protocol and standardize basic knowledge regarding the breathing technique, all participants will receive an initial educational session delivered on the first day of the on-site intervention. This session will include an introductory lecture and an explanatory leaflet outlining the fundamental principles of functional breathing and its relevance to the intervention.
  Interventions: Other: Therapeutic exercise + initial education session

INTERVENTIONS:
Other: Controlled breathing exercise protocol + therapeutic exercise + initial education session — In addition to the therapeutic exercise protocol and the educational session on proper breathing, participants will perform a controlled breathing protocol at home twice daily, at least five days per week, throughout the 6-week study period, following the recommendations of the principal investigator. The goal is to integrate slow, gentle, diaphragmatic, nasal breathing into daily life. Additionally, within this same group, two in-person controlled breathing training sessions, each lasting 5 minutes, will be conducted at the hospital to promote correct execution of the technique, one at the beginning of the intervention and another at its completion.
  To promote adherence and ensure correct and consistent execution, participants will have access through the Web-App to two audio files containing guided breathing instructions and visualization exercises. These recordings were specifically developed for this project by a physiotherapist with more than 20 years of experience.
  Arms: Therapeutic exercise + initial education session + home-based controlled breathing exercise protocol
Other: Therapeutic exercise + initial education session — In addition to the educational session on proper breathing, participants will perform:
  * Three weekly sessions of mobility and muscle-strengthening exercises (two on-site and one home-based) for 6 weeks. The on-site sessions will last between 30 and 40 minutes and will take place at the Rehabilitation Department of Hospital 12 de Octubre in Madrid (a total of 12 on-site sessions-two per week). The home-based exercise program will consist of completing, once per week during the 6-week intervention, a structured session that replicates the logic and technique of the on-site program. A maximum of four absences from the on-site therapeutic exercise program will be allowed, and on those occasions the patient must register via the web application that they completed the prescribed home-based program.
  * Walk a minimum of 7,000 steps/day or 50 minutes/day, three days per week.
  Arms: Therapeutic exercise + initial educational session on proper breathing

SUMMARY:
A randomized, parallel, double-blind, controlled, clinical trial. Two groups of participants will be included, both receiving a therapeutic exercise intervention and an educational session on the importance of proper breathing over a 6-week period. One of the groups will additionally perform a home-based controlled breathing exercise protocol. Pre- and post-intervention assessments (6 weeks) will be conducted, along with a follow-up evaluation 4 weeks after completion of the intervention. The goal is to determine the effectiveness of adding a controlled breathing exercise program to a therapeutic exercise intervention on cardiorespiratory variables in individuals with multiple myeloma.

DETAILED DESCRIPTION:
Randomized, parallel, double-blind, controlled clinical trial including participants with a confirmed medical diagnosis of multiple myeloma who are currently receiving active treatment with daratumumab and are under clinical follow-up by the Hospital Hematology Department.

Participants will be randomly assigned to one of two intervention groups:

* Control group: Therapeutic exercise + an initial educational session on proper breathing.
* Experimental group: Therapeutic exercise + an initial educational session on proper breathing + a home-based controlled breathing exercise protocol.

Both groups will undergo their respective intervention programs for 6 weeks. During each of the six weeks, participants will:

Perform three weekly sessions of mobility and muscle-strengthening exercises (two supervised on-site sessions and one home-based session). The on-site sessions will last 30-40 minutes and will be conducted at the Rehabilitation Department of Hospital 12 de Octubre in Madrid (a total of 12 on-site sessions, two per week). The weekly home-based session will consist of a structured session replicating the content and methodology of the supervised program.

Walk a minimum of 7,000 steps per day or 50 minutes per day, at least three days per week.

Participants assigned to the experimental group will additionally perform a controlled breathing protocol twice daily at home, following the recommendations of the principal investigator. Furthermore, they will complete two in-person controlled breathing training sessions, each lasting 5 minutes, at the hospital to ensure correct execution of the technique-one at the beginning of the intervention and one at its completion.

The variables to be assessed will include heart rate variability (HRV) indicators (SDNN, RMSSD, HF), heart rate, lower limb strength assessed using the 30-Second Sit-to-Stand Test (30STS), and estimated peak oxygen consumption (VO₂peak). All outcome measures will be evaluated at baseline, at the end of the 6-week intervention, and 4 weeks after completion of the intervention.

In addition, heart rate variability indicators and heart rate will be assessed immediately before and after the two in-person controlled breathing training sessions. as well as before and after an additional reinforcement session conducted four weeks after completion of the intervention. This will allow evaluation of the acute response of these variables to the breathing protocol, compared with participants in the control group, who will be instructed to breathe spontaneously, maintaining their habitual breathing pattern without any external guidance during the same time period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Confirmed diagnosis of multiple myeloma, currently undergoing active treatment with daratumumab, and under clinical follow-up by the Hematology Department of HU12O.
* Explicit medical indication for supervised physical activity issued by the responsible hematologist and documented in the medical record.
* No scheduled hematopoietic stem cell transplantation within the 60 days following the planned start date of the intervention (verified through medical record review).
* Functional status of ECOG 0-2 (Eastern Cooperative Oncology Group), assessed by a healthcare professional from the Hematology Department, ensuring the ability to perform at least basic and light instrumental activities of daily living, including independent ambulation.
* Access to a smartphone with stable internet connection, required for monitoring and recording adherence to the intervention.
* Ability to provide written informed consent, demonstrating understanding of the study's nature, purpose, and procedures.

Exclusion Criteria:

* Medical risk contraindicating exercise or breathing techniques:

  * Clinically significant cardiovascular disease, including:decompensated heart failure, acute myocardial infarction within the past 3 months, clinically uncontrolled arrhythmias, unstable angina, acute-phase deep vein thrombosis or pulmonary embolism, pacemakers or cardiac devices whose monitoring parameters contraindicate supervised exercise according to cardiology.
  * Severe decompensated respiratory disease, such as acute exacerbation of COPD, severe respiratory insufficiency, or persistently low resting oxygen saturation < 90% (not correctable).
* High musculoskeletal or bone risk:

  * Extensive lytic bone lesions, high risk of pathological fracture, or unstable vertebral fracture, documented by imaging or based on the assessment of the Hematology/Traumatology specialist.
  * Uncontrolled pain that prevents safe participation in an exercise program.
* Hematologic or systemic conditions contraindicating exercise:

  * Severe anemia: hemoglobin < 9 g/dL in women or < 8 g/dL in men (latest laboratory test ≤ 14 days).
  * Active systemic infection contraindicating exercise, fever ≥ 38 °C, or neutropenia < 0.5 × 10⁹/L.
  * Severe cytopenias that, in the opinion of the hematologist, preclude moderate exercise.
* Functional or procedural limitations:

  * Inability to remain in the supine position for ≥ 5 minutes, required for part of the breathing intervention.
  * Confirmed pregnancy or reasonable suspicion of pregnancy.
  * Severe cognitive impairment, major psychiatric disorders, or neurological diseases that limit understanding of the procedures or safe participation.
  * Significant difficulty understanding the language (spoken or written) that prevents following essential instructions or completing validated questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
HRV SDNN pre-postintervention | Baseline measurement: obtained prior to initiation of the training protocol. Second measurement: obtained immediately upon completion of the 6-week protocol.Follow-up: one additional measurement four weeks after completing the intervention protocol.
  Two measurement systems will be used concurrently to assess HRV SDNN and to evaluate agreement between methods:
  * Handheld portable electrocardiograph.
  * Heart rate and HRV monitor with chest-worn sensor (Polar H10).

SECONDARY OUTCOMES:
HRV SDNN In-person controlled breathing intervention | -First measurement: before and after the first in-person breathing training session.-Second measurement (week 6): before and after the second in-person breathing training session.-Third measurement (week 10): before and after the reinforcement session
  The standard deviation of normal R-R intervals (SDNN) is a heart rate variability (HRV) index that represents overall HRV activity in the time domain; higher values indicate greater overall HRV activity.
  This variable will be assessed before and after the two in-person 5-minute controlled breathing training sessions, as well as before and after an additional reinforcement session conducted four weeks after completion of the intervention. This design will allow evaluation of the temporal evolution of these variables in response to the breathing protocol, compared with participants in the control group, who will be instructed during the same time periods to breathe spontaneously, maintaining their usual breathing pattern without any external guidance.
  Two measurement systems will be used concurrently to assess HRV SDNN and to evaluate agreement between methods:
  * Handheld portable electrocardiograph.
  * Heart rate and HRV monitor with chest-worn sensor (Polar H10).
HRV RMSSD In-person controlled breathing intervention | -First measurement: before and after the first in-person breathing training session.-Second measurement (week 6): before and after the second in-person breathing training session.-Third measurement (week 10): before and after the reinforcement session.
  The root mean square of successive differences between R-R intervals (RMSSD) is a heart rate variability (HRV) index that correlates with vagally mediated regulation.
  This variable will be assessed before and after the two in-person 5-minute controlled breathing training sessions, as well as before and after an additional reinforcement session conducted four weeks after completion of the intervention. This design will allow evaluation of the temporal evolution of these variables in response to the breathing protocol, compared with participants in the control group, who will be instructed during the same time periods to breathe spontaneously, maintaining their usual breathing pattern without any external guidance.
  Two measurement systems will be used concurrently to assess HRV RMSSD and to evaluate agreement between methods:
  * Handheld portable electrocardiograph.
  * Heart rate and HRV monitor with chest-worn sensor (Polar H10).
HRV HF In-person controlled breathing intervention | -First measurement: before and after the first in-person breathing training session.-Second measurement (week 6): before and after the second in-person breathing training session.-Third measurement (week 10): before and after the reinforcement session.
  High frequency (HF) is a heart rate variability (HRV) index that represents parasympathetic nervous system activity in the frequency domain.
  This variable will be assessed before and after the two in-person 5-minute controlled breathing training sessions, as well as before and after an additional reinforcement session conducted four weeks after completion of the intervention. This design will allow evaluation of the temporal evolution of these variables in response to the breathing protocol, compared with participants in the control group, who will be instructed during the same time periods to breathe spontaneously, maintaining their usual breathing pattern without any external guidance.
  Two measurement systems will be used concurrently to assess HRV HF and to evaluate agreement between methods:
  * Handheld portable electrocardiograph.
  * Heart rate and HRV monitor with chest-worn sensor (Polar H10).
Heart Rate In-person controlled breathing intervention | -First measurement: before and after the first in-person breathing training session.-Second measurement (week 6): before and after the second in-person breathing training session.-Third measurement (week 10): before and after the reinforcement session.
  This variable will be assessed before and after the two in-person 5-minute controlled breathing training sessions, as well as before and after an additional reinforcement session conducted four weeks after completion of the intervention. This design will allow evaluation of the temporal evolution of these variables in response to the breathing protocol, compared with participants in the control group, who will be instructed during the same time periods to breathe spontaneously, maintaining their usual breathing pattern without any external guidance.
  Two measurement systems will be used concurrently to assess HR and to evaluate agreement between methods. Heart rate (HR) will be assessed using the mean value obtained over the 5-minute recording period from both measurement systems employed. These two systems are:
  * Handheld portable electrocardiograph.
  * Heart rate and HRV monitor with chest-worn sensor (Polar H10).
Heart Rate pre-postintervention | Baseline measurement: obtained prior to initiation of the training protocol. Second measurement: obtained immediately upon completion of the 6-week protocol.Follow-up: one additional measurement four weeks after completing the intervention protocol.
  Heart rate (HR) will be assessed using the mean value obtained over the 5-minute recording period from both measurement systems employed. These two systems are:
  * Handheld portable electrocardiograph.
  * Heart rate and HRV monitor with chest-worn sensor (Polar H10).
HRV RMSSD pre-postintervention | Baseline measurement: obtained prior to initiation of the training protocol. Second measurement: obtained immediately upon completion of the 6-week protocol.Follow-up: one additional measurement four weeks after completing the intervention protocol.
  The root mean square of successive differences between R-R intervals (RMSSD) is a heart rate variability (HRV) index that correlates with vagally mediated regulation. Two measurement systems will be used concurrently to assess HRV RMSSD and to evaluate agreement between methods:
  * Handheld portable electrocardiograph.
  * Heart rate and HRV monitor with chest-worn sensor (Polar H10).
HRV HF pre-postintervention | Baseline measurement: obtained prior to initiation of the training protocol. Second measurement: obtained immediately upon completion of the 6-week protocol.Follow-up: one additional measurement four weeks after completing the intervention protocol.
  High frequency (HF) is a heart rate variability (HRV) index that represents parasympathetic nervous system activity in the frequency domain; lower values indicate anxiety or stress, whereas higher values suggest a state of relaxation. Two measurement systems will be used concurrently to assess HRV HF and to evaluate agreement between methods:
  * Handheld portable electrocardiograph.
  * Heart rate and HRV monitor with chest-worn sensor (Polar H10).

OTHER OUTCOMES:
Lower-Limb Strength | Information for this variable will be collected at three time points: at baseline, at the end of the intervention (6 weeks), and four weeks after completion of the protocol.
  The 30-Second Sit-to-Stand test (30STS) will be used to assess lower-limb strength and endurance. This test has been employed in several studies involving oncology patients.
Estimated Peak Oxygen Consumption (VO₂peak) | Information for this variable will be collected at three time points: at baseline, at the end of the intervention (6 weeks), and four weeks after completion of the protocol.
  The same test used to assess lower-limb muscle strength (30STS) will be employed to estimate peak oxygen consumption (VO₂peak). The 30STS has been shown to be a useful tool for estimating VO₂peak in patients with cancer. Its use may facilitate the evaluation and stratification of functional capacity in this population. The formula used to estimate VO₂peak will correspond to the equation known as ONCORE.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Plaza-Manzano, PhD, Study Director — Faculty of Nursing, Physiotherapy and Podiatry. Universidad Complutense de Madrid

REFERENCES:
- [Background] Díaz-Balboa E, González-Salvado V, Rodríguez-Romero B, et al. Thirty-second sit-to-stand test as an alternative for estimating peak oxygen uptake and 6-min walking distance in women with breast cancer: a cross-sectional study. Support Care Cancer. 2022;30(10):8251-8260. doi:10.1007/s00520-022-07268-z
- [Background] Insulander P, Carnlöf C, Schenck-Gustafsson K, Jensen-Urstad M. Device profile of the Coala Heart Monitor for remote monitoring of the heart rhythm: overview of its efficacy. Expert Rev Med Devices. 2020;17(3):159-165. doi:10.1080/17434440.2020.1732814
- [Background] Luna-Alcala S, Espejel-Guzmán A, Lerma C, et al. Heart rate variability-based prediction of early cardiotoxicity in breast-cancer patients treated with anthracyclines and trastuzumab. Cardiooncology. 2024;10(1):32. doi:10.1186/s40959-024-00236-y
- [Background] Li J, Peng Y, Zhan D, Zhang Y, Yu S. Exercise interventions in patients with multiple myeloma: a scoping review. BMC Sports Sci Med Rehabil. 2025 Jun 9;17(1):148. doi: 10.1186/s13102-025-01193-4. PMID 40490782
- [Background] Nicol JL, Chong JE, McQuilten ZK, Mollee P, Hill MM, Skinner TL. Safety, Feasibility, and Efficacy of Exercise Interventions for People With Multiple Myeloma: A Systematic Review. Clin Lymphoma Myeloma Leuk. 2023 Feb;23(2):86-96. doi: 10.1016/j.clml.2022.10.003. Epub 2022 Oct 22. PMID 36450625
- [Background] Fournie C, Verkindt C, Dalleau G, Bouscaren N, Mohr C, Zunic P, Cabrera Q. Rehabilitation program combining physical exercise and heart rate variability biofeedback in hematologic patients: a feasibility study. Support Care Cancer. 2022 Mar;30(3):2009-2016. doi: 10.1007/s00520-021-06601-2. Epub 2021 Oct 12. PMID 34636946
- [Background] Shahriari M, Dehghan M, Pahlavanzadeh S, Hazini A. Effects of progressive muscle relaxation, guided imagery and deep diaphragmatic breathing on quality of life in elderly with breast or prostate cancer. J Educ Health Promot. 2017 Apr 19;6:1. doi: 10.4103/jehp.jehp_147_14. eCollection 2017. PMID 28546966